CLINICAL TRIAL: NCT00934544
Title: A Randomized Study of Ruxolitinib Tablets Compared to Best Available Therapy in Subjects With Primary Myelofibrosis, Post-Polycythemia Vera-Myelofibrosis or Post-Essential Thrombocythemia Myelofibrosis
Brief Title: Controlled Myelofibrosis Study With Oral Janus-associated Kinase (JAK) Inhibitor Treatment-II: The COMFORT-II Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CINC424A2352; CINCB 18424-352 (Other: INCYTE); 2009-009858-24 (EudraCT Number)
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Results first posted 2012-05-30 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Post-Essential Thrombocythemia Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- Ruxolitinib (Experimental): 5 mg tablets administered orally in an outpatient setting according to the protocol-specified dosing schedule
  Interventions: Drug: Ruxolitinib
- Best Available Therapy (BAT) (Active Comparator): Commercially available therapy, oral or parenteral, per manufacturer's instructions and Investigator discretion. BAT included the option of no treatment.
  Patients randomized to BAT were eligible to cross over to receive open-label ruxolitinib after a qualifying progression event, if they met the safety criteria. After the primary analysis in January 2011, patients randomized to receive BAT were allowed to cross over to receive ruxolitinib and move to the extension phase of the study without a qualifying progression event.
  Interventions: Drug: Best Available Therapy (BAT)

INTERVENTIONS:
Drug: Ruxolitinib — 5 mg tablets packaged as 60-count in high-density polyethylene bottles
  Arms: Ruxolitinib
Drug: Best Available Therapy (BAT) — Prescribing and usage per respective package inserts
  Arms: Best Available Therapy (BAT)

SUMMARY:
This was an open label, randomized study comparing the efficacy and safety of randomized 2:1 Ruxolitinib tablets versus best-available therapy, as selected by the investigator. The purpose was to compare the efficacy, safety and tolerability of Ruxolitinib (INC424/INCB018424) given twice daily to the best-available therapy, in subjects with primary myelofibrosis (PMF), post polycythemia vera myelofibrosis (PPV-MF) or post essential thrombocythemia myelofibrosis (PET-MF).

DETAILED DESCRIPTION:
This study included a randomized treatment phase, followed by an extension phase. The treatment phase lasted from Study Day 1 (day of randomization) to the occurrence of a protocol-specified progressive disease event or study conclusion, whichever came first. The extension phase (including crossover of control group patients) lasted from the progressive disease event until the earliest of the following events: a) the patient was no longer receiving clinical benefit, b) the patient chose to withdraw from the study, or c) the study ended. All patients received ruxolitinib in the extension phase of the study. Maximum individual patient duration was 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be diagnosed with PMF, PPV-MF or PET-MF according to the 2008 World Health Organization criteria
* Subjects with MF requiring therapy must be classified as high risk OR intermediate risk level 2 according to the prognostic factors defined by the International Working Group
* Subjects with an ECOG performance status of 0, 1, 2 or 3
* Subjects with peripheral blood blast count of < 10%.
* Subjects who have not previously received treatment with a JAK inhibitor

Exclusion Criteria:

* Subjects with a life expectancy of less than 6 months
* Subjects with inadequate bone marrow reserve as demonstrated by specific clinical laboratory counts
* Subjects with any history of platelet counts < 50,000/µL or ANC < 500/µL except during treatment for a myeloproliferative disorder or treatment with cytotoxic therapy for any other reason
* Subjects with inadequate liver or renal function
* Subjects with clinically significant bacterial, fungal, parasitic or viral infection which require therapy
* Subjects with an active malignancy over the previous 5 years except specific skin cancers
* Subjects with severe cardiac conditions
* Subjects who have had splenic irradiation within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2015-03-04 (Actual); Study Completion 2015-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (58):
- Austria (4):
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (9):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, La Louvière
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Roeselare
  - Novartis Investigative Site, Yvoir
- France (15):
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lens
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (9):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Frankfurt/M
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
- Italy (6):
  - Novartis Investigative Site, Pavia, (PV)
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Orbassano
  - Novartis Investigative Site, Pavia
- Netherlands (6):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, The Hague
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Valencia, Valencia
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Stockholm
- United Kingdom (4):
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Oxford

REFERENCES:
- [Derived] Verstovsek S, Gotlib J, Mesa RA, Vannucchi AM, Kiladjian JJ, Cervantes F, Harrison CN, Paquette R, Sun W, Naim A, Langmuir P, Dong T, Gopalakrishna P, Gupta V. Long-term survival in patients treated with ruxolitinib for myelofibrosis: COMFORT-I and -II pooled analyses. J Hematol Oncol. 2017 Sep 29;10(1):156. doi: 10.1186/s13045-017-0527-7. PMID 28962635
- [Derived] McMullin MF, Harrison CN, Niederwieser D, Demuynck H, Jakel N, Gopalakrishna P, McQuitty M, Stalbovskaya V, Recher C, Theunissen K, Gisslinger H, Kiladjian JJ, Al-Ali HK. The use of erythropoiesis-stimulating agents with ruxolitinib in patients with myelofibrosis in COMFORT-II: an open-label, phase 3 study assessing efficacy and safety of ruxolitinib versus best available therapy in the treatment of myelofibrosis. Exp Hematol Oncol. 2015 Sep 15;4:26. doi: 10.1186/s40164-015-0021-2. eCollection 2015. PMID 26380150
- [Derived] Vannucchi AM, Kantarjian HM, Kiladjian JJ, Gotlib J, Cervantes F, Mesa RA, Sarlis NJ, Peng W, Sandor V, Gopalakrishna P, Hmissi A, Stalbovskaya V, Gupta V, Harrison C, Verstovsek S; COMFORT Investigators. A pooled analysis of overall survival in COMFORT-I and COMFORT-II, 2 randomized phase III trials of ruxolitinib for the treatment of myelofibrosis. Haematologica. 2015 Sep;100(9):1139-45. doi: 10.3324/haematol.2014.119545. Epub 2015 Jun 11. PMID 26069290
- [Derived] Cervantes F, Vannucchi AM, Kiladjian JJ, Al-Ali HK, Sirulnik A, Stalbovskaya V, McQuitty M, Hunter DS, Levy RS, Passamonti F, Barbui T, Barosi G, Harrison CN, Knoops L, Gisslinger H; COMFORT-II investigators. Three-year efficacy, safety, and survival findings from COMFORT-II, a phase 3 study comparing ruxolitinib with best available therapy for myelofibrosis. Blood. 2013 Dec 12;122(25):4047-53. doi: 10.1182/blood-2013-02-485888. Epub 2013 Oct 30. PMID 24174625
- [Derived] Wilkins BS, Radia D, Woodley C, Farhi SE, Keohane C, Harrison CN. Resolution of bone marrow fibrosis in a patient receiving JAK1/JAK2 inhibitor treatment with ruxolitinib. Haematologica. 2013 Dec;98(12):1872-6. doi: 10.3324/haematol.2013.095109. Epub 2013 Sep 20. PMID 24056820
- [Derived] Mesa RA, Kiladjian JJ, Verstovsek S, Al-Ali HK, Gotlib J, Gisslinger H, Levy R, Siulnik A, Gupta V, Khan M, DiPersio JF, McQuitty M, Catalano JV, Hunter DS, Knoops L, Deininger M, Cervantes F, Miller C, Vannucchi AM, Silver RT, Barbui T, Talpaz M, Barosi G, Winton EF, Mendeson E, Harvey JH Jr, Arcasoy MO, Hexner E, Lyons RM, Paquette R, Raza A, Sun W, Sandor V, Kantarjian HM, Harrison C. Comparison of placebo and best available therapy for the treatment of myelofibrosis in the phase 3 COMFORT studies. Haematologica. 2014 Feb;99(2):292-8. doi: 10.3324/haematol.2013.087650. Epub 2013 Aug 2. PMID 23911705
- [Derived] Harrison C, Kiladjian JJ, Al-Ali HK, Gisslinger H, Waltzman R, Stalbovskaya V, McQuitty M, Hunter DS, Levy R, Knoops L, Cervantes F, Vannucchi AM, Barbui T, Barosi G. JAK inhibition with ruxolitinib versus best available therapy for myelofibrosis. N Engl J Med. 2012 Mar 1;366(9):787-98. doi: 10.1056/NEJMoa1110556. PMID 22375970

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 9 countries located in Europe: Austria, Belgium, France, Germany, Italy, Netherlands, Spain, Sweden, and United Kingdom.
Pre-assignment Details: 219 unique participants were randomized to either ruxolitinib or BAT. Of the 73 participants randomized to BAT, 45 were crossed over to ruxolitinib after a protocol-specified qualifying disease progression event.
Groups:
- Ruxolitinib; Ruxolitinib After BAT (Cross-over): 5 milligram tablets administered orally in an outpatient setting according to the protocol-specified dosing schedule
- Best Available Therapy (BAT): Commercially available therapy, oral or parenteral, per manufacturer's instructions and Investigator discretion. BAT included the option of no treatment.
Period: Primary Endpoint Analysis (Interim)
Arm/Group | Ruxolitinib | Best Available Therapy (BAT) | Ruxolitinib After BAT (Cross-over)
Started | 146 | 73 | 0
Completed | 91 | 31 | 0
Not Completed | 55 | 42 | 0
Not completed — Adverse Event | 12 | 4 | 0
Not completed — Withdrawal by Subject | 2 | 9 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Disease Progression | 1 | 3 | 0
Not completed — Non-compliance with study Medication | 2 | 0 | 0
Not completed — Non-compliance with study procedures | 0 | 1 | 0
Not completed — Other reasons | 7 | 7 | 0
Not completed — Entered extension phase | 29 | 18 | 0
Period: Overall Disposition at 5 Year Follow-up
Arm/Group | Ruxolitinib | Best Available Therapy (BAT) | Ruxolitinib After BAT (Cross-over)
Started | 146 | 28 | 45
Crossed Over After Qualifying Event | 0 | 0 | 27
Crossed Over After AMEND 5 | 0 | 0 | 12
Crossed Over: Other | 0 | 0 | 6
Completed | 39 | 0 | 11
Not Completed | 107 | 28 | 34
Not completed — Including stem cell transplantation | 16 | 9 | 6
Not completed — Adverse Event | 35 | 5 | 10
Not completed — Withdrawal by Subject | 10 | 9 | 0
Not completed — Protocol Violation | 2 | 0 | 5
Not completed — Disease progression | 32 | 4 | 7
Not completed — Noncompliance with study medication | 4 | 0 | 1
Not completed — Noncompliance with study procedures | 0 | 1 | 0
Not completed — Lack of Efficacy | 8 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib | Best Available Therapy (BAT) | Total
Number analyzed (Participants) | 146 | 73 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (9.74) | 65.2 (10.27) | 65.2 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 31 | 94
  Male | 83 | 42 | 125
Disease Profile - Type of Myelofibrosis (MF) [Count of Participants; unit: Participants] — Disease characteristics at baseline. Overall, (primary myelofibrosis (PMF), post-polycythemia vera-myelofibrosis(PPV-MF) and post-essential thrombocythemia-myelofibrosis (PET-MF) were diagnose in participants. The frequency of PMF was similar between ruxolitinib and BAT arms. In addition, the frequencies of PPV-MF and PET-MF were also similar between both treatment arms.
  Participants
    Primary Myelofibrosis | 77 | 39 | 116
    Post-polycythemia vera-myelofibrosis | 48 | 20 | 68
    Post-essential thrombocythemia-myelofibrosis | 21 | 14 | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 35% Reduction in Spleen Volume From Baseline at Week 48
Description: The change in spleen volume from baseline to week 48 was measured by magnetic resonance imaging (MRI) (or by computer tomography (CT) for participants unable to undergo MRI) and was calculated only for participants who had an evaluable spleen volume at baseline. The percentage of participants achieving a greater than or equal to 35% reduction in spleen volume from baseline to week 48 was then calculated by treatment group.
Time Frame: Baseline, Week 48
Population: Full analysis set (FAS) consisted of all subjects who were randomized and put in strata according to International Working Group for Myelofibrosis Research and Treatment(IWG MRT) prognostic criteria. The table included participants with non-missing baseline MRI measurement of spleen volume only.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 144 | 72
Percentage of Participants | 28.5 | 0
Statistical Analysis 1: Comparison: Ruxolitinib vs Best Available Therapy (BAT); Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Kaplan-Meir estimate = 28.1, 95% CI 2-sided [21.3 to 36.6], Standard Deviation 22.123

2. Secondary Outcome: Duration of Maintenance of Spleen Volume Reduction (Median)
Description: DoMSR is defined as the interval between the first spleen volume measurement that is >=35% reduction from baseline and the first scan that is no longer = 35% reduction AND that is a >25% increase over nadir. It was evaluated using the Kaplan-Meier estimate for each treatment arm. The analysis was performed only for subjects who achieved greater than 35% reduction in spleen volume.
Time Frame: Baseline, up to Year 5
Population: Full analysis set (FAS) consisted of all subjects who were randomized and put in strata according to International Working Group for Myelofibrosis Research and Treatment(IWG MRT) prognostic criteria. Treatment groups were defined according to the treatment assignment at the time of randomization.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 78 | 1
years | 3.22 [1.65 to NA] — Upper limit is not estimable | NA [NA to NA] — There was only one BAT patient responder (≥ 35% reduction in spleen volume) but no consecutive readings to determine any value for duration of response - no Median or CI possible to calculate

3. Secondary Outcome: Duration of Maintenance of Spleen Volume Reduction (Kaplan-Meier Estimates)
Description: This is defined as the interval between randomization and date of the first MRI showing a 35% reduction from baseline in spleen volume. The analysis was performed for participants who achieved a 35% reduction in spleen volume.
Time Frame: Baseline, up to Year 5
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: probability of response
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 78 | 1
probability of response
  1.0 year | 0.72 [.60 to .81] | NA [NA to NA] — There was only one BAT patient responder (≥ 35% reduction in spleen volume) but no consecutive readings to determine any value for duration of response - no Median or CI possible to calculate
  1.5 years | 0.67 [0.55 to 0.77] | NA [NA to NA] — There was only one BAT patient responder (≥ 35% reduction in spleen volume) but no consecutive readings to determine any value for duration of response - no Median or CI possible to calculate
  2.0 years | 0.63 [0.50 to 0.73] | NA [NA to NA] — There was only one BAT patient responder (≥ 35% reduction in spleen volume) but no consecutive readings to determine any value for duration of response - no Median or CI possible to calculate
  2.5 years | 0.54 [0.41 to 0.65] | NA [NA to NA] — There was only one BAT patient responder (≥ 35% reduction in spleen volume) but no consecutive readings to determine any value for duration of response - no Median or CI possible to calculate
  3.0 years | 0.51 [0.38 to 0.62] | NA [NA to NA] — There was only one BAT patient responder (≥ 35% reduction in spleen volume) but no consecutive readings to determine any value for duration of response - no Median or CI possible to calculate
  3.5 years | 0.48 [0.35 to 0.60] | NA [NA to NA] — There was only one BAT patient responder (≥ 35% reduction in spleen volume) but no consecutive readings to determine any value for duration of response - no Median or CI possible to calculate
  4.0 years | 0.48 [0.35 to 0.60] | NA [NA to NA] — There was only one BAT patient responder (≥ 35% reduction in spleen volume) but no consecutive readings to determine any value for duration of response - no Median or CI possible to calculate
  4.5 years | 0.48 [0.35 to 0.60] | NA [NA to NA] — There was only one BAT patient responder (≥ 35% reduction in spleen volume) but no consecutive readings to determine any value for duration of response - no Median or CI possible to calculate
  5.0 years | 0.48 [0.35 to 0.60] | NA [NA to NA] — There was only one BAT patient responder (≥ 35% reduction in spleen volume) but no consecutive readings to determine any value for duration of response - no Median or CI possible to calculate

4. Secondary Outcome: Percentage of Participants With at Least 35% Reduction in Spleen Volume From Baseline at Week 24
Description: The change in spleen volume from baseline to week 24 was measured by magnetic resonance imaging (MRI) (or by computer tomography (CT) for participants unable to undergo MRI) and was calculated only for participants who had an evaluable spleen volume at baseline. The percentage of participants achieving a greater than or equal to 35% reduction in spleen volume from baseline to week 24 was then calculated by treatment group.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 144 | 72
Percentage of Participants | 31.9 | 0

5. Secondary Outcome: Time to First at Least 35% Reduction in Spleen Volume From Baseline by Treatment (Primary Analysis)
Description: This is defined as the interval between randomization and date of the first MRI showing at least 35% reduction from baseline in spleen volume. The analysis was performed for participants who achieved a 35% reduction in spleen volume
Time Frame: Time from randomization and date of the first MRI showing at least 35% reduction from baseline in spleen volume
Population: Full analysis set (FAS)
Measure: Number (95% Confidence Interval); unit: probability of response
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 69 | 1
probability of response
  12 weeks | 0.23 [0.14 to 0.34] | 0 [NA to NA] — There was only one BAT patient responder (≥ 35% reduction in spleen volume) but no consecutive readings to determine any value for duration of response - no Median or CI possible to calculate
  24 weeks | 0.67 [0.54 to 0.76] | 1 [NA to NA] — There was only one BAT patient responder (≥ 35% reduction in spleen volume) but no consecutive readings to determine any value for duration of response - no Median or CI possible to calculate
  36 weeks | 0.87 [0.76 to 0.93] | 1 [NA to NA] — There was only one BAT patient responder (≥ 35% reduction in spleen volume) but no consecutive readings to determine any value for duration of response - no Median or CI possible to calculate
  48 weeks | 0.97 [0.89 to 0.99] | 1 [NA to NA] — There was only one BAT patient responder (≥ 35% reduction in spleen volume) but no consecutive readings to determine any value for duration of response - no Median or CI possible to calculate

6. Secondary Outcome: Progression-free Survival (PFS)
Description: Median of time progression free survival (95% CI), years
Time Frame: Time from randomization and the earliest of either increase in spleen volume >=25% from on-study nadir, splenic irradiation, splenectomy, leukemic transformation or death
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 146 | 73
years | 1.6 [1.2 to 2.3] | 1.4 [1.1 to 1.9]

7. Secondary Outcome: Leukemia-free Survival (LFS)
Description: Time from randomization and earliest of either (1) date of bone marrow blast count of 20% or greater; (2) date of first peripheral blast count of 20% or greater that was subsequently confirmed to sustain for at least 8 weeks; (3) date of death from any cause
Time Frame: Time from randomization and earliest of either leukemia or death
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 146 | 73
Years | NA [NA to NA] — Values are not estimable as Median was not reached | 4.1 [2.4 to NA] — Upper limit was not estimable

8. Secondary Outcome: Overall Survival (OS)
Description: Defined as the interval between randomization and the date of the bone marrow blast count of 20% or greater OR the date of the first peripheral blast count of 20% or greater that was subsequently confirmed to have been sustained for at least 8 weeks OR the date of death from any cause, whichever occurs first. OS was summarized using Kaplan-Meier estimates for each treatment arm. The estimates were supplemented by tables of number of events and probability estimates at several timepoints
Time Frame: From randomization until death from any cause
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Years
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 146 | 73
Years | NA [NA to NA] — Values are not estimable as Median was not reached | 4.1 [2.4 to NA] — Upper limit of CI was not estimable

9. Secondary Outcome: Percentage of Participants With Bone Marrow Histomorphology at Week 48 (Primary Analysis)
Description: This was noted as fibrosis density and was tabulated by fibrosis grade at baseline and at week 48 (post-baseline). Descriptive statistics (participant percentages) were used.
  Fibrosis grades: 0 Scattered linear reticulin with no intersections corresponding to normal bone marrow ; 1 Loose network of reticulin with many intersections, especially in perivascular areas; 2 Diffuse and dense increase in reticulin with extensive intersections, occasionally with only focal bundles of collagen and/or focal osteosclerosis; 3 Diffuse and dense increase in reticulin with extensive intersections with coarse bundles of collagen, often associated with significant osteosclerosis
Time Frame: 48 weeks
Population: Full analysis set (FAS) consisted of all subjects who were randomized and put in strata according to International Working Group for Myelofibrosis Research and Treatment(IWG MRT) prognostic criteria.
Measure: Number; unit: Percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 146 | 73
Percentage of participants
  Grade 0 | 2.7 | 0.0
  Grade 1 | 7.5 | 2.7
  Grade 2 | 8.9 | 6.8
  Grade 3 | 24.0 | 15.1
  Missing Grade | 56.8 | 75.3

10. Secondary Outcome: Bone Marrow Histomorphology
Description: Shift table from baseline to last available postbaseline fibrosis grade by treatment
  The grade gives an indication of the activity or amount of inflammation and the stage represents the amount of fibrosis or scarring. The grade is assigned a number based on the degree of inflammation, which is usually scored from 0-4 with 0 being no activity and 3 or 4 considered severe activity
Time Frame: Baseline, once a year
Population: Full Analysis Set (FAS)
  Numbers of Participants Analyzed reflect only those participants who were randomized to either Ruxolitinib or Best Available Therapy and do not count those participants who could have crossed over to Ruxolitinib
Measure: Number; unit: participants
Arm/Group | Ruxolitinib | Ruxolitinib - Grade 1 | Ruxolitinib - Grade 2 | Ruxolitinib - Grade 3 | Ruxolitinib - Missing | Best Available Therapy (BAT) - Grade 0 | Best Available Therapy (BAT) - Grade 1 | Best Available Therapy (BAT) - Grade 2 | Best Available Therapy (BAT) - Grade 3 | Best Available Therapy - Missing
Number analyzed (Participants) | 146 | 146 | 146 | 146 | 146 | 73 | 73 | 73 | 73 | 73
participants
  Postbaseline Grade 0 | 1 [41.8 to 2.3] | 1 [47.9 to 1.9] | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0
  Postbaseline Grade 1 | 0 | 10 | 9 | 2 | 0 | 0 | 1 | 0 | 1 | 0
  Postbaseline Grade 2 | 0 | 2 | 8 | 8 | 1 | 0 | 0 | 4 | 1 | 0
  Postbaseline Grade 3 | 0 | 6 | 19 | 28 | 2 | 0 | 0 | 4 | 8 | 3
  Postbaseline Missing | 2 | 2 | 17 | 20 | 3 | 2 | 2 | 19 | 24 | 4

11. Secondary Outcome: Duration of Follow-up by Treatment
Description: Number of Participants with duration of Follow up
Time Frame: baseline, 260 weeks (end of study)
Population: Safety Set
  Numbers of Participants Analyzed reflect only those participants who were randomized to either Ruxolitinib or Best Available Therapy and do not count those participants who could have crossed over to Ruxolitinib
Measure: Number; unit: participants
Arm/Group | Ruxolitinib | Best Available Therapy (BAT)
Number analyzed (Participants) | 146 | 73
participants
  <=1 year | 16 | 15
  >1 year - <=2 years | 21 | 10
  >2 years - <=3 years | 9 | 13
  >3 years - <=4 years | 12 | 5
  >4 years - <=5 years | 27 | 8
  5 years | 61 | 22

ADVERSE EVENTS:
Groups:
- Ruxolitinib Randomized: Ruxolitinib Randomized
- Ruxolitinib Randomized + Extension Phase: Ruxolitinib Randomized + Extension Phase
- BAT Randomized: BAT Randomized
- Ruxolitinib Cross-over: Ruxolitinib cross-over
Arm/Group | Ruxolitinib Randomized | Ruxolitinib Randomized + Extension Phase | BAT Randomized | Ruxolitinib Cross-over
Serious Adverse Events (participants affected / at risk) | 51/146 | 85/146 | 22/73 | 20/45
Other Adverse Events (participants affected / at risk) | 145/146 | 145/146 | 64/73 | 42/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib Randomized (N=146) | Ruxolitinib Randomized + Extension Phase (N=146) | BAT Randomized (N=73) | Ruxolitinib Cross-over (N=45)
Anaemia (Blood and lymphatic system disorders) | 8 | 10 | 4 | 2
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0
Paratracheal lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 2 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 4
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 2 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 4 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 3 | 5 | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 3 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Keratitis (Eye disorders) | 1 | 1 | 0 | 0
Ocular vascular disorder (Eye disorders) | 1 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 6 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric varices (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 3 | 4 | 0 | 1
Asthenia (General disorders) | 1 | 1 | 1 | 0
Chest pain (General disorders) | 1 | 2 | 0 | 0
Disease progression (General disorders) | 1 | 1 | 0 | 0
General physical health deterioration (General disorders) | 2 | 4 | 1 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1
Performance status decreased (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 4 | 5 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 2 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 2 | 1 | 0
Bronchitis (Infections and infestations) | 3 | 4 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 1 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Febrile infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 3 | 0 | 0
Gastroenteritis clostridial (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0
Genital infection female (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 3 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 2 | 2 | 0 | 0
Meningitis (Infections and infestations) | 1 | 1 | 0 | 0
Meningoencephalitis herpetic (Infections and infestations) | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Oesophageal infection (Infections and infestations) | 0 | 1 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 2 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 11 | 4 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 1 | 0 | 0
Postoperative abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 3 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0 | 1
Sepsis syndrome (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 2 | 0 | 1
Skin infection (Infections and infestations) | 1 | 2 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Testicular abscess (Infections and infestations) | 1 | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 2 | 2 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 3 | 0 | 0
Viral infection (Infections and infestations) | 1 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ear injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 1 | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 2 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 4 | 0 | 0
Coma (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 0
Pseudoradicular syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 3 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 2 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 4 | 1 | 3
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal infarct (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0
Aortic thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Arterial stenosis (Vascular disorders) | 1 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 1 | 0 | 0
Intra-abdominal haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib Randomized (N=146) | Ruxolitinib Randomized + Extension Phase (N=146) | BAT Randomized (N=73) | Ruxolitinib Cross-over (N=45)
Anaemia (Blood and lymphatic system disorders) | 61 | 71 | 8 | 19
Leukocytosis (Blood and lymphatic system disorders) | 7 | 8 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 67 | 77 | 10 | 21
Angina pectoris (Cardiac disorders) | 5 | 8 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 11 | 1 | 1
Palpitations (Cardiac disorders) | 8 | 12 | 0 | 2
Tachycardia (Cardiac disorders) | 4 | 8 | 4 | 1
Vertigo (Ear and labyrinth disorders) | 5 | 9 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 7 | 11 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 14 | 21 | 12 | 3
Abdominal pain upper (Gastrointestinal disorders) | 12 | 16 | 4 | 5
Ascites (Gastrointestinal disorders) | 4 | 6 | 3 | 3
Constipation (Gastrointestinal disorders) | 12 | 19 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 36 | 55 | 13 | 12
Dyspepsia (Gastrointestinal disorders) | 7 | 10 | 4 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 10 | 0 | 2
Nausea (Gastrointestinal disorders) | 21 | 30 | 7 | 5
Vomiting (Gastrointestinal disorders) | 16 | 27 | 1 | 4
Asthenia (General disorders) | 28 | 38 | 9 | 10
Chest pain (General disorders) | 0 | 0 | 4 | 4
Chills (General disorders) | 4 | 8 | 0 | 0
Fatigue (General disorders) | 23 | 36 | 8 | 8
General physical health deterioration (General disorders) | 3 | 7 | 4 | 3
Oedema peripheral (General disorders) | 33 | 55 | 21 | 8
Peripheral swelling (General disorders) | 3 | 7 | 0 | 3
Pyrexia (General disorders) | 20 | 36 | 6 | 7
Bronchitis (Infections and infestations) | 15 | 37 | 5 | 3
Cystitis (Infections and infestations) | 9 | 15 | 3 | 1
Gastroenteritis (Infections and infestations) | 9 | 14 | 1 | 1
Herpes zoster (Infections and infestations) | 9 | 16 | 0 | 5
Lower respiratory tract infection (Infections and infestations) | 2 | 2 | 0 | 3
Nasopharyngitis (Infections and infestations) | 27 | 40 | 9 | 4
Respiratory tract infection (Infections and infestations) | 6 | 9 | 3 | 2
Rhinitis (Infections and infestations) | 7 | 9 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 9 | 1 | 2
Urinary tract infection (Infections and infestations) | 11 | 19 | 2 | 6
Fall (Injury, poisoning and procedural complications) | 4 | 8 | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 3 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 3 | 3 | 0 | 3
Cardiac murmur (Investigations) | 6 | 8 | 3 | 3
Gamma-glutamyltransferase increased (Investigations) | 7 | 11 | 1 | 1
Haemoglobin decreased (Investigations) | 4 | 6 | 3 | 4
Platelet count decreased (Investigations) | 11 | 12 | 2 | 9
Weight decreased (Investigations) | 3 | 8 | 6 | 2
Weight increased (Investigations) | 23 | 29 | 1 | 5
White blood cell count increased (Investigations) | 3 | 4 | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 6 | 20 | 4 | 4
Gout (Metabolism and nutrition disorders) | 1 | 6 | 1 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 8 | 1 | 0
Iron overload (Metabolism and nutrition disorders) | 2 | 5 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 30 | 8 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 24 | 10 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 9 | 4 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 28 | 5 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 8 | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 11 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 9 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 24 | 4 | 11
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 11 | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 10 | 1 | 0
Dizziness (Nervous system disorders) | 12 | 20 | 5 | 6
Headache (Nervous system disorders) | 18 | 23 | 4 | 8
Paraesthesia (Nervous system disorders) | 10 | 16 | 4 | 4
Sciatica (Nervous system disorders) | 5 | 9 | 1 | 0
Anxiety (Psychiatric disorders) | 5 | 9 | 0 | 1
Insomnia (Psychiatric disorders) | 9 | 13 | 7 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 38 | 12 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 35 | 13 | 12
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 11 | 13 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 18 | 5 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 3 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 1 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 | 8 | 0 | 4
Eczema (Skin and subcutaneous tissue disorders) | 1 | 3 | 4 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 11 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 14 | 27 | 6 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 17 | 13 | 4
Rash (Skin and subcutaneous tissue disorders) | 8 | 12 | 1 | 2
Rosacea (Skin and subcutaneous tissue disorders) | 2 | 4 | 1 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 12 | 0 | 2
Haematoma (Vascular disorders) | 15 | 22 | 3 | 4
Hypertension (Vascular disorders) | 8 | 19 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.